CLINICAL TRIAL: NCT02878941
Title: Synovial Fluid Analysis of Intraarticular Elbow Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00072559
Record Dates: First submitted 2016-07-13; First posted 2016-08-25 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-01

CONDITIONS: Elbow Fracture; Joint Contracture
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elbow Fracture (Other): Patients with an intraarticular elbow fracture and/or dislocation. Synovial fluid from the injured elbow will be obtained during the subject's emergency department encounter by one of the Chief Residents or Attending surgeon as part of standard of care procedures for pain control-related injection and aspiration. Patients with an intraarticular elbow fracture and/or dislocation receive an intraarticular elbow injection with anesthetic (i.e. lidocaine or marcaine) to provide analgesia for elbow range of motion testing and orthopaedic reduction maneveuers as the current standard of care. The patients would be asked to consent for 2 elbow joint aspirations: 1.Aspiration of the injured elbow at time of surgical fracture fixation; 2.Aspiration of the uninjured elbow at time of surgical fracture fixation.
  Interventions: Procedure: Synovial Fluid Analysis

INTERVENTIONS:
Procedure: Synovial Fluid Analysis — Synovial fluid aspiration (act of using an 18 gauge needle to obtain synovial fluid from the elbow) in the emergency room for patients with the eligible elbow fracture (as defined in inclusion/exclusion criteria) is performed in conjunction with the anesthetic injection as part of standard of care. The elbow will be prepped as per usual for the anesthetic injection. An 18 gauge needle will be inserted through a lateral approach. The subject's elbow will be aspirated. The syringe with the aspirate would be removed from the needle while the needle would remain in the subject's elbow joint. The syringe with anesthetic would then be connected to the needle, and the anesthetic would be injected into the elbow joint. Therefore, no risks from a separate aspiration would be conferred to the patient.

SUMMARY:
The objective of this study is to obtain and compare bilateral elbow joint synovial fluid from patients with unilateral intraarticular elbow fracture and a contralateral healthy appearing elbow joint. The synovial fluid samples will undergo several forms of analysis for metabolites and proteins. Matched-pair statistical analysis will be performed to determine the metabolites and proteins that may play the greatest role in development of joint contracture.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Intraarticular elbow fracture (humerus, radial head and/or ulna fracture)

Exclusion Criteria:

* Age <18 years
* Open elbow fracture
* Bilateral elbow fractures
* Patients with history of osteomyelitis of elbow
* Inflammatory arthropathy (ie. Rheumatoid arthritis)
* Prior surgery on fractured elbow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
metabolite composition of synovial fluid | time of fracture until surgical fixation (up to 5 weeks after injury)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided